CLINICAL TRIAL: NCT05560698
Title: A Motivation-enhancing Intervention to Retain Participants in a Trial After Treatment With Allergen Immunotherapy
Brief Title: A Motivation-enhancing App to Retain Patients With Hay Fever in a Trial After Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other); Innovation Fund Denmark (Individual)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 26092022
Record Dates: First submitted 2022-09-21; First posted 2022-09-29 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2023-11

CONDITIONS: Grass Pollen Allergy; Rhinoconjunctivitis
Keywords: Retention; Motivation; Self-Determination Theory; Grass Pollen Allergic Rhinoconjunctivitis; Intralymphatic Immunotherapy; Patient and Public Involvement

STUDY DESIGN:
Intervention Model Description: Participants are randomized 1:1 across treatment group
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Other): Standard reporting method
  Interventions: Other: Standard intervention
- Intervention (Other): Web based motivation-enhancing app
  Interventions: Other: Motivation-enhancing intervention

INTERVENTIONS:
Other: Motivation-enhancing intervention — The web app is designed as an efficient and easy-to-use app configurable to personal preferences. Each day participants receive a text message on their smartphone with a link for the daily cSMS questionnaire. The questionnaire addresses the same questions as the questionnaire in the standard intervention, but the format is different, and some shortcuts makes it easier to answer. When the questionnaire is answered, the web app gives access to different features. The following features distinct the motivation-enhancing intervention from the standard intervention (1) only complete the entire questionnaire on days with symptoms, (2) integration of grass pollen counts and forecasts, (3) showing personal response rate, (4) access to own data via a graph, (5) advice against grass pollen allergy, (6) status of the study, (7) individually choosing the time of response, (8) option to download an icon for the home screen and (9) contact information. The development is an ongoing iterative process
  Arms: Intervention
Other: Standard intervention — Each day participants receive a text message on their smartphone with a link for the daily cSMS questionnaire. When the questionnaire is answered, the tab needs to be closed.
  Arms: Control

SUMMARY:
The motivation-enhancing intervention is designed for participants in the ILIT.NU trial. The participants are patients with hay fever who are treated with a vaccination in an inguinal lymph node. The motivation-enhancing intervention is a web-based app developed in collaboration with patient partners and is intended to increase retention and reporting in the ILIT.NU trial.

DETAILED DESCRIPTION:
The ILIT.NU trial (EudraCT 2020-001060-28) investigates whether patient reported outcome measures compound symptom-medication score (cSMS) are relieved by intralymphatic immunotherapy (ILIT). The participants are asked for a three-year period to attend annual consultations and to daily fill in an online questionnaire about their allergy symptoms and medication use during the grass pollen season (100 days).

High attrition rates have been a problem in previous ILIT trials. High attrition affects generalizability, validity and reliability of a trial. To increase retention and reporting in the ILIT.NU trial, a motivation-enhancing web-based app has been developed. The web app is based on the Self-Determination Theory and is developed in collaboration with patient partners and clinicians. Participants are randomized across treatment group to either the motivation-enhancing web app or the standard reporting method. The project is conducted as a Study Within a Trial (SWAT).

ELIGIBILITY:
Inclusion Criteria:

* Participants enrolled in the ILIT.NU trial

Exclusion Criteria:

* Participants not enrolled in the ILIT.NU trial, Denmark

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2022-09-26 (Actual); Primary Completion 2023-08-17 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Rate of reporting daily cSMS data | 16 weeks
  Increased reporting will be compared within and between the intervention group and the control group, to evaluate the effectiveness of the motivation-enhancing intervention

SECONDARY OUTCOMES:
Retention | 16 weeks
  Increased retention measured as loss to follow up, where drop outs from the ILIT.NU trial will be compared within and between the intervention group and the control group, to evaluate the effectiveness of the motivation-enhancing intervention
Motivation | 14 days
  Increased motivation measured by the Intrinsic Motivation Inventory Questionnaire, to evaluate the effectiveness of the motivation-enhancing intervention
Participant experience with the web-based app | 12 weeks
  10 participants are invited to a focus group interview to discuss their experiences with the web-based app

CONTACTS AND LOCATIONS:
Overall Officials: Anne Poder Petersen, Principal Investigator — University of Aarhus
Locations (1):
- Anne Poder Petersen, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No
Due to restrictions from GDPR and the Danish National Committee on Health Research Ethics, IPD are not shared with other researchers. Anonymous data may be shared.

REFERENCES:
- See also: Home page for the ILIT.NU trial — http://ilit.nu